CLINICAL TRIAL: NCT00278655
Title: Hematopoietic Stem Cell Therapy for Patients With Inflammatory Multiple Sclerosis Failing Interferon Therapy: A Phase II Multi-Center Trial
Brief Title: Hematopoietic Stem Cell Therapy for Patients With Multiple Sclerosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAD MS.Auto2002
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hematopoietic stem cell transplantation (Experimental): All participants will undergo hematopoietic stem cell transplantation after receiving conditioning regimen.
  Interventions: Biological: Hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: Hematopoietic stem cell transplantation — Autologous hematopoietic stem cell transplantation

SUMMARY:
Multiple sclerosis is disease believed to be due to immune cells, cells which normally protect the body, but are now attacking the tissue in the brain and possibly the spinal cord. The likelihood of progression of this disease is high. This study is designed to examine whether treating patients with high dose cyclophosphamide and CAMPATH-1H (drugs which reduce the function of the immune system) followed by return of previously collected blood stem cells will stop the progression of your multiple sclerosis. Stem cells are undeveloped cells that have the capacity to grow into mature blood cells, which normally circulate in the blood stream. The purpose of the cyclophosphamide and CAMPATH-1H is to destroy the cells in your immune system which are thought to be causing your disease. The purpose of the stem cell infusion is to restore the body's blood production, which will be severely impaired by the high dose chemotherapy and to produce a normal immune system that will no longer attack the body.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-50, inclusive.
2. Diagnosis of Multiple Sclerosis (MS) using Poser criteria (Appendix A).
3. An Expanded Disability Status Scale (EDSS) of 2.0 - 5.5 (Appendix B).
4. Inflammatory disease despite primary disease modifying therapy with at least 3 months of interferon. Failure is defined as two or more clinical relapses with documented neurologic changes within the year prior to the study. (NOTE: Relapses must have required treatment with corticosteroids. Sensory only relapses are excluded.) Failure may also be defined as one relapse within the year prior to study if there is evidence on MRI of active inflammation (i.e., gadolinium enhancement).

Exclusion Criteria:

1. Any illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive chemotherapy.
2. Prior history of malignancy except localized basal cell, squamous skin cancer or carcinoma in situ of the cervix. Other malignancies for which the patient is judged to be cured, such as head and neck cancer, or breast cancer will be considered on an individual basis.
3. Positive pregnancy test.
4. Inability or unwillingness to pursue effective means of birth control. Effective birth control is defined as 1) refraining from all acts of vaginal intercourse (ABSTINENCE); 2) consistent use of birth control pills; 3) injectable birth control methods (Depo-provera, Norplant); 4) tubal sterilization or male partner who has undergone vasectomy; 5) placement of an intrauterine device (IUD); or 6) use, with every act of intercourse, of diaphragm with contraceptive jelly and/or condoms with contraceptive foam.
5. Failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
6. Forced expiratory volume in 1 second (FEV1) / forced vital capacity (FVC) < 60% of predicted after bronchodilator therapy (if necessary).
7. Diffusing capacity of the lung for carbon monoxide (DLCO) < 50% of predicted.
8. Resting left ventricular ejection fraction (LVEF) < 50 %.
9. Bilirubin > 2.0 mg/dl.
10. Serum creatinine > 2.0 mg/dl.
11. Known hypersensitivity to mouse, rabbit, or E. Coli derived proteins, or to iron compounds/medications.
12. Presence of metallic objects implanted in the body that would preclude the ability of the patient to safely have MRI exams.
13. Diagnosis of primary progressive multipole sclerosis (MS).
14. Platelet count < 100,000/ul.
15. Psychiatric illness, mental deficiency or cognitive dysfunction making compliance with treatment or informed consent impossible.
16. Active infection except asymptomatic bacteruria.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2003-06; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2003 and February 2005 in Northwestern Memorial Hospital 21 patients with relapsing-remitting multiple sclerosis (MS) underwent autologous hematopoietic stem cell transplantation in order to evaluate the safety and clinical outcome of autologous non-myeloablative hematopoetic stem cell transplantation in MS.
Pre-assignment Details: 21 eligible patients had relapsing remitting MS not responding to interferon and had had two corticosteroid -treated relapses within the previous 12 months or one relapse and gadolinium-enhancing lesions seen on MRI and separate from the relapse.
Groups:
- Autologous Hematopoietic Stem Cell Transplantation: Patient's own blood stem cells collected after mobilization with cyclophosphamide (2.0 gm/m²)and granulocyte colony-stimulating factor (G-CSF) (5-10mcg/kg/day.Collected stem cells given back to the patient after receiving conditioning regimen (Cyclophosphamide 50 mg/kg/day for four days and either 20 mg alemtuzumab or 6mg/kg rabbit antithymocyte globulin.
Period: Overall Study
Arm/Group | Autologous Hematopoietic Stem Cell Transplantation
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Stem Cell Transplantation: All participants will undergo stem cell transplantation after receiving conditioning regimen.
  hematopoietic stem cell transplantation : Autologous hematopoietic stem cell transplantation
Arm/Group | Stem Cell Transplantation
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Disease Progression
Description: Data are reporting number of participants with disease progression. Disease progression is defined as a 1 point increase in the Expanded Disability Status Scale (EDSS) on consecutive evaluations at least 3 months apart.
Time Frame: 3 years after transplant
Measure: Number; unit: participants
Groups:
- Stem Cell Transplantation: Autologous hematopoietic stem cell transplantation Peripheral blood stem cells were mobilised with 2g per square m intravenous (IV) cyclophosphamide (CY) followed by 10 µg per kg subcutaneous filgrastim daily from day 5. After neutrophil recovery, the mobilised cells were collected by apheresis. The recovered cells were unselected and cryopreserved. There was at least three weeks between mobilisation and the conditioning regimen. The conditioning regimen used was 200 mg per kg intravenous CY , given in four equal fractions between day -5 and day -2 with IV mesna, and one 20mg dose of IV alemtuzumab (CAMPATH-1H) given on day -2 with 250 mg intravenous methyl-prednisolone as premedication. Alemtuzumab was changed to rabbit antithymocyte globulin rATG) in the last 4 patients, who received 6 mg per kg rATG over 5 days instead of alemtuzumab . Stem cells wer reinfused 36 h after completion of CY. 5 µg/kg/day filgrastim was given from day 5 until neutrophil recovery.
Arm/Group | Stem Cell Transplantation
Number analyzed (Participants) | 21
participants | 4

2. Secondary Outcome: Survival
Description: Data are reporting the number of participants who survived three years after the transplant
  Survival of 21 participants was evaluated at three years after the transplant
Time Frame: three years
Measure: Number; unit: participants
Groups:
- Autologous Hematopoietic Stem Cell Transplantation: Patient's own blood stem cells collected after mobilization with cyclophosphamide (2.0 gm/m²)and G-CSF (5-10 mcg/kg/day.Collected stem cells given back to the patient after receiving conditioning regimen (Cyclophosphamide 50 mg/kg/day for four days and either 20 mg alemtuzumab or 6mg/kg rabbit antithymocyte globulin.
Arm/Group | Autologous Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 21
participants | 21

ADVERSE EVENTS:
Time Frame: three years
Arm/Group | Stem Cell Transplantation
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 7/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Transplantation (N=21)
Transient neurological symptoms (Nervous system disorders) | 1 (1) — One patient had Transient neurological symptoms that manifested as leftsided hypoaesthesia, which was attributed to a filgrastim-related flair. The neurological symptoms resolved when the drug was discontinued.
Blood culture with coagulase-negative staphylococcus (Infections and infestations) | 1 (1) — One patient had a blood culture with coagulase-negative staphylococcus; this was isolated in one specimen of four sent concurrently, which suggests a probable contaminant.
Dermatomal zoster (Infections and infestations) | 2 (2) — Two patients developed dermatomal zoster at 20 and 22 months post-transplantation and both resolved with oral antiviral therapy.
Diarrhoea due to Clostridium difficile (Gastrointestinal disorders) | 1 (1) — One month after hospital discharge after the transplantation, one patient developed diarrhoea due to Clostridium difficile that resolved with oral metronidazole.
Grade IV thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) — Two patients treated with alemtuzumab developed grade IV thrombocytopenia 7 and 14 months after transplantation. The thrombocytopenia presented as easy bruising and petechiae, resolved with intravenous immunoglobulin, prednisone and rituximab

LIMITATIONS AND CAVEATS:
The study had following limitations: small number of enrolled participants and no randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No